CLINICAL TRIAL: NCT01851447
Title: Pilot Study to Assess Biomarkers of Changes in Barrier Function of Skeletal Muscle in Patients With a Fragile Sarcolemmal Muscular Dystrophy
Brief Title: Skeletal Muscle Biomarkers in People With Fragile Sarcolemmal Muscular Dystrophy
Status: Active, not recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health Clinical Center (CC) (NIH); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130112; 13-CH-0112
Record Dates: First submitted 2013-05-09; First posted 2013-05-10 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2025-07-16

CONDITIONS: Genetic Disorder
Keywords: Membrane Wound; Inflammatory Cytokines; Exercise; Plasma Membrane Repair; Predictors of Outcome; Natural History
MeSH Terms: conditions — Genetic Diseases, Inborn; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fragile Sarcolemmal Muscular Dystrophy: patients with early adulthood or late onset of a genetic disorder FSMD (LGMD 2B-F, I, L, MM, BMD and MMD3)

SUMMARY:
Background:

- Some kinds of muscular dystrophy affect the skeletal muscle membrane. In these conditions, the muscle membrane is more fragile. This affects how the muscles contract and relax, which causes movement problems. Researchers are looking at several muscle enzymes, or chemicals that affect how muscle cells function. By studying changes in these enzymes, they may be able to better understand how muscular dystrophy affects the cells. Researchers want to collect biomarkers (chemicals from blood samples) from people with fragile sarcolemmal muscular dystrophy. This information may provide better treatments for this condition.

Objectives:

- To study biomarkers that may affect the muscles of people with fragile sarcolemmal muscular dystrophy.

Eligibility:

- Individuals at least 18 years of age with fragile sarcolemmal muscular dystrophy.

Design:

* Participants will be screened with a medical history and physical exam.
* Participants will be asked to come for four visits to the National Institutes of Health Clinical Center. The visits will be at least 2 months apart. Each visit will require participants to stay for 5 days at the clinical center.
* During each visit, participants will provide frequent small blood samples. These samples will be collected while at rest and after physical exercise.
* Participants will also have a physical therapy assessment. They will perform standard motor function tests and imaging tests (MRI, MRS). These tests may take up to 1 hour each time.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Objectives: the aim of this protocol is to identify biomarker and clinical correlates of changes in the barrier function of skeletal muscle membrane (i.e. cell membrane permeability) before and after routine motor function testing in patients with one of the Fragile Sarcolemmal Muscular Dystrophies (FSMD).

Study population: patients with early adulthood or later onset of a FSMD (LGMD2B-F, I, L, MM, BMD, and MMD3).

Study Phase: pilot study. Outcome measures: increased change in baseline levels of proteins that are released into the blood from damaged skeletal muscle, such as Creatine Kinase (CK), Lactate Dehydrogenase (LDH), Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), troponins, and myoglobin in plasma, changes in inflammation markers, circulating microRNAs and imaging studies to identify effective biomarkers for use in future clinical trials.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Aged 18 or older
* Have a confirmed genetic diagnosis of one of the FSMDs or have a clinical phenotype consistent with one of the FSMDs
* Be able to travel to the NIH Clinical Center at the NIH for studies
* Able to commit to multiple 5 day stays at the NIH Clinical Center
* Established primary care physician
* Ambulant: able to walk 10 meters or 33 feet without walking aids or orthotics

EXCLUSION CRITERIA:

* Fail to meet the above inclusion criteria
* Are unable or unwilling to be examined
* Adults unable to provide their own consent
* Have active, on-going medical problems such as (e.g. diabetes, hypothyroidism, pancreatitis, anemia, cancer, renal, hepatic, pulmonary or cardiac disease) or who have undergone recent surgery (i.e. less than 8 days post-surgery)
* Pregnant females
* Currently taking any or a combination of anti-inflammatory drugs, statins or other drugs with known myotoxicity, narcotics

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 11 patients, 18 years or older with early adulthood or later onset of a genetically diagnosed FSMD will be enrolled in this study. We estimate no more than 50 patients to be eligible for enrollment. This pilot study will accept a maximum of 11 patients.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in biomarker levels | early in the morning, before and after morning activities
  biomarker levels (CK, ALT, AST...) increases
changes in biomarker levels | after physical exercise, strength test under guidance of physical therapist
  biomarker levels (CK, ALT, AST...) increase

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Zimmerberg, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-CH-0112.html